CLINICAL TRIAL: NCT02874508
Title: Association of Circulating Leukocyte Subpopulations and Cardio Vascular Events in the Perioperative Period
Brief Title: Leukocytes and Perioperative Cardio Vascular Events
Acronym: LeukoCAPE
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Johann Motsch, Prof. Dr., University Hospital Heidelberg
Other Study IDs: LeukoKAPE01
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Elective Non-cardiac Surgery
Keywords: leukocyte subpopulations; perioperative myocardial infarction; non-cardiac surgery; perioperative cardiovascular risk

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
To analyze whether non-cardiac surgery in high-risk cardio-vascular patients induces a quantitative change in one or several leukocyte subpopulations and whether such changes are associated with perioperative cardio-vascular events.

DETAILED DESCRIPTION:
Annually, there are more than 200 million surgeries worldwide (Weiser et al., 2016; Weiser et al., 2008). The POISE study revealed 5% of patients undergoing a non-cardiac surgery suffer perioperative myocardial infarcts going along with a perioperative mortality rate of about 11,6% (Devereaux et al., 2011). Possibilities to preoperatively identify patients at risk are limited (Devereaux und Sessler, 2015; Gillmann et al., 2014) and prophylactic interventions are not yet established or controversial (Devereaux und Sessler, 2015).

Selected leukocyte subpopulations have been demonstrated to be associated with higher risk for cardiovascular events (Berg et al., 2012; Cheng et al., 2008; Engelbertsen et al., 2012; Kotfis et al., 2015; Rogacev et al., 2011; Rogacev et al., 2012).The aim of this study is to analyze whether surgical stress (non-cardiac surgery) induces a quantitative change in one or several of these leukocyte subpopulations and whether quantitative changes are associated with perioperative cardiovascular events. Therefore, high-risk cardio-vascular patients scheduled for non-cardiac surgery will be recruited. Blood will be drawn at predefined time points before surgery and up to three days postoperatively. Leukocytes will be analyzed by flow cytometry. During 30 day follow up adverse cardiovascular events will be recorded. ECGs will be recorded preoperatively and on post-OP day 3. High-sensitive cardiac Troponin T will be measured prior to the operation and on post-OP day one to three. The patient chart will be screened for cardio vascular events up to day 30. A telephone interview will be performed to detect cardiovascular events after discharge until post-OP day 30.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Coronary heart disease
* Non-cardiac surgery
* Inpatient treatment
* Informed consent

Exclusion Criteria:

* 17 years of age or younger
* Known pregnancy or breastfeeding
* Missing informed consent
* Ambulatory or day-case surgery
* Emergency surgery
* Acute or chronic leukemia
* Current leukocytosis
* Current aplasia or leukopenia
* Current GM-CSF treatment
* Carotid artery surgery
* History of splenectomy or indications of splenectomy
* Cortisone treatment within past 14 days
* History of organ transplantation
* Current immunosuppressive medication
* Chemotherapy completed less than 14 days ago
* Intraoperative dexamethasone application
* Entity which is part of the composite endpoint diagnosed within past 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to University Hospital Heidelberg suffering coronary heart disease and scheduled for non-cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Composite Endpoint | 30 days postoperative
  Composite of: cardiac death, myocardial ischemia, myocardial infarction, embolic or thrombotic stroke, congestive heart failure, serious cardiac arrhythmia

SECONDARY OUTCOMES:
Individual components of the composite endpoint | 30 days postoperative
Peripheral vascular occlusion | 30 days postoperative
New onset atrial fibrillation | 30 days postoperative
Acute kidney injury | 30 days postoperative
Myocardial injury after non-cardiac surgery | 30 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Johann Motsch, Prof. Dr., Principal Investigator — Department of Anethesiology, University Hospital Heidelberg
Locations (1):
- Department of Anesthesiology, University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogacev KS, Cremers B, Zawada AM, Seiler S, Binder N, Ege P, Grosse-Dunker G, Heisel I, Hornof F, Jeken J, Rebling NM, Ulrich C, Scheller B, Bohm M, Fliser D, Heine GH. CD14++CD16+ monocytes independently predict cardiovascular events: a cohort study of 951 patients referred for elective coronary angiography. J Am Coll Cardiol. 2012 Oct 16;60(16):1512-20. doi: 10.1016/j.jacc.2012.07.019. Epub 2012 Sep 19. PMID 22999728
- [Background] Berg KE, Ljungcrantz I, Andersson L, Bryngelsson C, Hedblad B, Fredrikson GN, Nilsson J, Bjorkbacka H. Elevated CD14++CD16- monocytes predict cardiovascular events. Circ Cardiovasc Genet. 2012 Feb 1;5(1):122-31. doi: 10.1161/CIRCGENETICS.111.960385. Epub 2012 Jan 11. PMID 22238190
- [Background] Devereaux PJ, Xavier D, Pogue J, Guyatt G, Sigamani A, Garutti I, Leslie K, Rao-Melacini P, Chrolavicius S, Yang H, Macdonald C, Avezum A, Lanthier L, Hu W, Yusuf S; POISE (PeriOperative ISchemic Evaluation) Investigators. Characteristics and short-term prognosis of perioperative myocardial infarction in patients undergoing noncardiac surgery: a cohort study. Ann Intern Med. 2011 Apr 19;154(8):523-8. doi: 10.7326/0003-4819-154-8-201104190-00003. PMID 21502650
- [Background] Devereaux PJ, Sessler DI. Cardiac Complications in Patients Undergoing Major Noncardiac Surgery. N Engl J Med. 2015 Dec 3;373(23):2258-69. doi: 10.1056/NEJMra1502824. No abstract available. PMID 26630144
- [Background] Engelbertsen D, Andersson L, Ljungcrantz I, Wigren M, Hedblad B, Nilsson J, Bjorkbacka H. T-helper 2 immunity is associated with reduced risk of myocardial infarction and stroke. Arterioscler Thromb Vasc Biol. 2013 Mar;33(3):637-44. doi: 10.1161/ATVBAHA.112.300871. Epub 2013 Jan 10. PMID 23307873
- [Background] Gillmann HJ, Meinders A, Grohennig A, Larmann J, Bunte C, Calmer S, Sahlmann B, Rustum S, Aper T, Lichtinghagen R, Koch A, Teebken OE, Theilmeier G. Perioperative levels and changes of high-sensitivity troponin T are associated with cardiovascular events in vascular surgery patients. Crit Care Med. 2014 Jun;42(6):1498-506. doi: 10.1097/CCM.0000000000000249. PMID 24584063
- [Background] Kotfis K, Biernawska J, Zegan-Baranska M, Zukowski M. Peripheral Blood Lymphocyte Subsets (CD4+, CD8+ T Cells, NK Cells) in Patients with Cardiovascular and Neurological Complications after Carotid Endarterectomy. Int J Mol Sci. 2015 May 4;16(5):10077-94. doi: 10.3390/ijms160510077. PMID 25946343
- [Background] Rogacev KS, Seiler S, Zawada AM, Reichart B, Herath E, Roth D, Ulrich C, Fliser D, Heine GH. CD14++CD16+ monocytes and cardiovascular outcome in patients with chronic kidney disease. Eur Heart J. 2011 Jan;32(1):84-92. doi: 10.1093/eurheartj/ehq371. Epub 2010 Oct 12. PMID 20943670
- [Background] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Background] Weiser TG, Haynes AB, Molina G, Lipsitz SR, Esquivel MM, Uribe-Leitz T, Fu R, Azad T, Chao TE, Berry WR, Gawande AA. Size and distribution of the global volume of surgery in 2012. Bull World Health Organ. 2016 Mar 1;94(3):201-209F. doi: 10.2471/BLT.15.159293. PMID 26966331
- [Derived] Larmann J, Handke J, Scholz AS, Dehne S, Arens C, Gillmann HJ, Uhle F, Motsch J, Weigand MA, Janssen H. Preoperative neutrophil to lymphocyte ratio and platelet to lymphocyte ratio are associated with major adverse cardiovascular and cerebrovascular events in coronary heart disease patients undergoing non-cardiac surgery. BMC Cardiovasc Disord. 2020 May 18;20(1):230. doi: 10.1186/s12872-020-01500-6. PMID 32423376